CLINICAL TRIAL: NCT00270855
Title: Exercise to Reduce Obesity in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3918-R; UL1RR031990 (NIH)
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus; Obesity; Paraplegia; Quadriplegia; Spinal Cord Injury
Keywords: Body Composition; Exercise; Glucose Tolerance; Insulin Sensitivity; Functional Electric Stimulation
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Paraplegia; Quadriplegia; Spinal Cord Injuries; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm Crank Ergometer (Other): Upper body Cycle ergometer Exercise: 10-minute warm up, 40 minutes @ 70%HRMax (50RPM), 10 minute cool down 5x/week x 16 weeks
  Interventions: Procedure: Arm Crank Ergometry
- FESLCE (Other): Functional Electrical Stimulation Leg Cycle Ergometer Exercise: 10-minute warm up, 40 minutes @ 70%HRMax (50RPM), 10 minute cool down 5x/week x 16 weeks
  Interventions: Procedure: FES Cycle Ergometer

INTERVENTIONS:
Procedure: Arm Crank Ergometry — Use of an upper body cycle to perform exercise. 10-minute warm up, 40 minutes @ 70%HRMax (50RPM), 10 minute cool down 5x/week x 16 weeks
  Arms: Arm Crank Ergometer
Procedure: FES Cycle Ergometer — Use of an FES cycle ergometer to perform exercise. 10-minute warm up, 40 minutes @ 70%HRMax (50RPM), 10 minute cool down 5x/week x 16 weeks
  Arms: FESLCE

SUMMARY:
The purpose of this proposal was to evaluate and compare the health benefits of using upper extremity exercise versus functional electrical stimulation for lower extremity exercise. It was our hypothesis that both Functional Electrical Stimulation Leg Cycle Ergometry (FES LCE) exercise and voluntary Arm Crank Ergometry (ACE) upper extremity exercise would increase whole body energy expenditure, thereby increasing muscle mass, insulin sensitivity, glucose effectiveness and improving lipid profiles in adults with paraplegia.

DETAILED DESCRIPTION:
Objective: Spinal cord injuries (SCI) predispose individuals to impaired fitness, obesity, glucose intolerance and insulin resistance, placing them at greater risk for diabetes, coronary artery disease, and upper extremity overuse syndrome as body weight increases. The specific objectives for the current proposal were to compare the impact of FES (functional electrical stimulation) lower extremity exercise versus upper extremity arm crank ergometry on energy metabolism, body composition and fat deposition, insulin sensitivity, glucose effectiveness, lower extremity bone mineral density and lipid profiles, in adults with complete paraplegia. Research Plan: A randomized, baseline-controlled, prospective, 16-week interventional trial was employed to assess the impact of FES LCE versus volitional arm crank ergometry exercise on energy metabolism, body composition and fat deposition, insulin sensitivity, glucose effectiveness, lower extremity bone mineral density and lipid profiles in adults with complete paraplegia. Methods: Twenty-four 18-65 y.o. individuals with motor complete T4-L2 SCI were assigned to either FES lower extremity exercise or upper extremity arm crank ergometry to compare impact on energy expenditure, obesity, and insulin sensitivity. Both groups were provided similar nutritional assessments and intervention. Exercise training consisted of five, 40-minute sessions at 70% maximal heart rate (HRmax) each week for a total of 16 weeks. Resting metabolic rate, exercise energy expenditure, body composition by DXA, insulin sensitivity, glucose effectiveness, lipid profiles, and lower extremity bone mineral density (BMD) were determined before and after 16-week exercise interventions.

ELIGIBILITY:
Inclusion Criteria:

Criteria for participation included men and women within the age range of 18-65 years old with BMI>25 kg/m2 who have had T4-L2 Motor-Complete (ASIA A&B) SCI for duration of greater than 12 months to ensure a homogenous sample.

Exclusion Criteria:

* persons who were unresponsive to surface neurostimulation
* had participated in an FES or ACE exercise (> 60 minutes/week) program within the past 3 months
* and those with known orthopedic limitations
* CAD
* diabetes mellitus (fasting glucose>126 or HgbA1c>7.0) or known family history
* hypothyroidism
* and/or renal disease were excluded from the study.
* Additionally, individuals with uncontrolled autonomic dysreflexia, recent (within 3 months) deep vein thrombosis, or pressure ulcers > Grade II were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Gater, MD PhD MS, Principal Investigator — Hunter Holmes McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm Crank Ergometer: Upper body Cycle ergometer
  Arm Crank Ergometry: Use of an upper body cycle to perform exercise.
- FESLCE: Functional Electrical Stimulation Cycle Ergometer for Lower body
  FES Cycle Ergometer: Use of an FES cycle ergometer to perform exercise
Period: Overall Study
Arm/Group | Arm Crank Ergometer | FESLCE
Started | 15 | 14
Completed | 7 | 6
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Arm Cycling Ergometer: Upper body Cycle ergometer
  Arm Crank Ergometry: Use of an upper body cycle to perform exercise.
- Total: Total of all reporting groups
Arm/Group | Arm Cycling Ergometer | FESLCE | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (10) | 39 (14) | 40.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 4 | 9
% Body Fat [Mean (Standard Deviation); unit: Percent Body Fat] | 38.9 (6.9) | 41.6 (7.1) | 40.75 (7.4)
Fat Mass (Kg) [Mean (Standard Deviation); unit: Kg] | 29.6 (6.4) | 33.4 (11.0) | 31.5 (8.7)
Fat-Free Mass (kg) [Mean (Standard Deviation); unit: Kg] | 49.6 (9.1) | 49.5 (11.2) | 49.55 (10.15)
Glucose Effectiveness (Sg) [Mean (Standard Deviation); unit: min^-1] | 0.023 (0.01) | 0.017 (0.01) | 0.02 (0.01)
Insulin Sensitivity (Si) [Mean (Standard Deviation); unit: μu/ml] | 3.0 (2.0) | 2.7 (2.0) | 2.85 (2)
Exercise Energy Expenditure (Kcal/session) [Mean (Standard Deviation); unit: Kcal/session] | 128.3 (35.4) | 80.7 (32.6) | 101 (34)
Resting Metabolic Rate [Mean (Standard Deviation); unit: Kcal/d] | 1442 (348) | 1710 (974) | 1565 (689)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 176 (29) | 167 (49) | 172 (38)
HDL-Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 35.7 (6.4) | 37.8 (8.3) | 36.7 (7.1)
Bone Mineral Density [Mean (Standard Deviation); unit: g/cm^2] | 1.138 (0.104) | 1.293 (0.135) | 1.209 (0.140)

OUTCOME MEASURES:

1. Primary Outcome: Change in % Body Fat
Description: Change in % Body Fat after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: Percent Body Fat
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
Percent Body Fat | -1.83 (2.72) | -1.68 (0.98)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group (i.e, baseline vs. post-intervention in ARE); Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group (i.e, baseline vs. post-intervention in FESLCE); Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

2. Primary Outcome: Change in Fat Mass
Description: Change in Fat Mass (Kg) after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: Baseline, 16 Weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
Kg | -1.84 (1.99) | -1.02 (2.55)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

3. Primary Outcome: Change in Fat-Free Mass
Description: Fat-Free Mass (kg). Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
Kg | 0.90 (3.49) | 1.86 (2.42)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p = 0.519, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

4. Primary Outcome: Change in Glucose Effectiveness (Sg)
Description: Change in Glucose Effectiveness (min^-1). Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: Baseline, 16-weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: min^-1
Groups:
- Arm Crank Ergometer: Upper body Cycle ergometer Exercise: 10-minute warm up, 40 minutes @ 70%HRMax (50RPM), 10 minute cool down 5x/week x 16 weeks
  Arm Crank Ergometry: Use of an upper body cycle to perform exercise.
- FESLCE: Functional Electrical Stimulation Leg Cycle Ergometer Exercise: 10-minute warm up, 40 minutes @ 70%HRMax (50RPM), 10 minute cool down 5x/week x 16 weeks
  FES Cycle Ergometer: Use of an FES cycle ergometer to perform exercise
Arm/Group | Arm Crank Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
min^-1 | 0.00 (0.02) | 0.01 (0.01)
Statistical Analysis 1: Comparison: Arm Crank Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p = 0.615, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

5. Primary Outcome: Change in Insulin Sensitivity (Si)
Description: Change in insulin sensitivity (min^-1). Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: Baseline, 16-weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Arm Crank Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
min^-1 | 10.1 (25.3) | 5.28 (12.4)
Statistical Analysis 1: Comparison: Arm Crank Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

6. Primary Outcome: %Body Fat Between Groups
Description: Comparison of %body fat between the ACE and FESLCE groups following the 16 week intervention.
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: Percent Body Fat
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
Percent Body Fat | 37.1 (5.6) | 39.9 (6.8)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; We evaluated differences in the above variable between the ACE and FESLCE following the the 16-week exercise intervention; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Fat Mass Between Groups
Description: Comparison of fat mass between the ACE and FESLCE groups following the 16 week intervention.
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
kg | 29.6 (6.4) | 33.4 (11.0)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Fat Free Mass Between Groups
Description: Comparison of fat free mass between the ACE and FESLCE groups following the 16 week intervention.
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
kg | 50.5 (10.4) | 51.3 (12.8)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Insulin Sensitivity (Si) Between Groups
Description: Comparison of Si between the ACE and FESLCE groups following the 16 week intervention.
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
min^-1 | 13.7 (0.02) | 8.4 (12.9)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Glucose Effectiveness (Sg) Between Groups
Description: Comparison of Sg between the ACE and FESLCE groups following the 16 week intervention.
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
min^-1 | .03 (0.009) | 0.02 (0.009)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Lower Limb Bone Mineral Density
Description: Change in lower limb bone mineral density after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: g*(cm^2)^-1
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
g*(cm^2)^-1 | 0.02 (0.03) | -0.01 (0.02)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

12. Secondary Outcome: Change in Lower Limb Bone Mineral Content
Description: Change in lower limb bone mineral content after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
grams | -0.07 (0.14) | -0.06 (0.09)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

13. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
mg/dL | -1.14 (22.6) | -12.33 (8.19)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

14. Secondary Outcome: Change in High Density Lipoprotein Cholesterol (HDL)
Description: Change in HDL after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
mg/dL | -2.29 (3.55) | 0.07 (2.63)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

15. Secondary Outcome: Change in Low Density Lipoprotein Cholesterol (LDL)
Description: Change in LDL after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
mg/dL | 0.14 (20.7) | 1.43 (24.3)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

16. Secondary Outcome: Change in Total Cholesterol (TC)
Description: Change in TC after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
mg/dL | -1.14 (22.6) | -12.33 (8.19)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

17. Secondary Outcome: Change in the Ratio of Total Cholesterol to High Density Lipoprotein Cholesterol (TC:HDL)
Description: Change in TC:HDL after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: Baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
Ratio | 0.24 (0.59) | -0.22 (0.79)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

18. Secondary Outcome: Lower Limb Bone Mineral Density Between Groups
Description: Comparison of Lower limb bone mineral density between the ACE and FESLCE groups following the 16 week intervention
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: g*(cm^2)^-1
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
g*(cm^2)^-1 | 1.15 (0.12) | 1.28 (0.12)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Lower Limb Bone Mineral Content Between Groups
Description: Comparison of Lower limb bone mineral content between the ACE and FESLCE groups following the 16 week intervention
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
grams | 3.37 (0.64) | 2.88 (0.55)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Triglycerides Between Groups
Description: Comparison of Triglycerides between the ACE and FESLCE groups following the 16 week intervention
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
mg/dL | 87.33 (46.7) | 103.6 (65.16)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: High Density Lipoprotein Cholesterol (HDL) Between Groups
Description: Comparison of HDL between the ACE and FESLCE groups following the 16 week intervention
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
mg/dL | 33.43 (5.1) | 37.8 (8.3)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney-u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Low Density Lipoprotein Cholesterol (LDL) Between Groups
Description: Comparison of LDL between the ACE and FESLCE groups following the 16 week intervention
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
mg/dL | 118.3 (32.2) | 107.3 (35.2)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Other — A Mann-Whitney U test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Total Cholesterol (TC) Between Groups
Description: Comparison of TC between the ACE and FESLCE groups following the 16 week intervention
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
mg/dL | 172.0 (28.6) | 163.7 (38.9)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — We used a Mann-Whitney U test; p > 0.05, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Ratio of Total Cholesterol to High Density Lipoprotein Cholesterol (TC:HDL) Between Groups
Description: Comparison of Ratio of Total Cholesterol to High Density Lipoprotein Cholesterol (TC:HDL) between the ACE and FESLCE groups following the 16 week intervention
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
Ratio | 5.3 (1.4) | 4.5 (1.4)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A mann-whitney u test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

25. Other Pre Specified Outcome: Change in Resting Metabolic Rate
Description: Change in resting metabolic rate after 16 week intervention. Change score was calculated as final value (i.e., post intervention variable) minus baseline value.
Time Frame: baseline, 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
kcal/day | -131.7 (393) | -322.0 (963)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer; We evaluated differences between baseline and following the 16-week exercise intervention in the ACE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: FESLCE; We evaluated differences between baseline and following the 16-week exercise intervention in the FESLCE group; Test type: Non-Inferiority or Equivalence — A Wilcoxon signed-rank test was performed; p > 0.05, t-test, 2 sided

26. Other Pre Specified Outcome: Resting Metabolic Rate Between Groups
Description: Comparison of resting metabolic rate between the ACE and FESLCE groups following the 16 week intervention
Time Frame: 16 weeks
Population: Two exercise groups consisted of an arm crank ergometry group and an FESLCE group.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Arm Cycling Ergometer | FESLCE
Number analyzed (Participants) | 7 | 6
kcal/day | 1309.06 (167.9) | 1387.8 (392.3)
Statistical Analysis 1: Comparison: Arm Cycling Ergometer vs FESLCE; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A Mann-Whitney U test was performed; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Arm Cycling Ergometer | FESLCE
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
The number of subjects that withdrew lead to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No